CLINICAL TRIAL: NCT02233478
Title: Dietary Protein in Pomegranate Ellagitannin Bioavailability
Brief Title: Comparing the Effect of Whey and Soy Protein on the Absorption of Pomegranate Polyphenols in the Human Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine and Chief Division of Clinical Nutrition, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-000905
Record Dates: First submitted 2014-08-15; First posted 2014-09-08 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Pomegranate polyphenols; Soy Protein; Ellagitannins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pomegranate Juice (Active Comparator): Subjects will be asked to take a dietary supplement on the day of intervention. Prior to intervention, subjects will be asked to avoid high-polyphenol foods, certain vitamins, minerals, herbs and dietary supplements for 4 days, dietary instruction will be provided. Blood samples will be taken at screen for safety labs. On study days 5, 13 and 21 a spot urine will be collected and a 7 hr serial blood draw will be performed at 0 hr, 30 min, 1 hr, 2 hr, 3 hr, 4 hr and 6 hr. Subjects will be provided with a light lunch with foods low in polyphenols. Subjects will only be able to eat the foods provided on the intervention days. Subjects will be asked to drink 32oz of water during the 7-hr period. Subjects will also be asked to collect all of their urines for 24 hrs, 2 consecutive days.
  Interventions: Dietary Supplement: Pomegranate Juice
- Soybean Flour Protein (Active Comparator): Subjects will be asked to take a dietary supplement on the day of intervention. Prior to intervention, subjects will be asked to avoid high-polyphenol foods, certain vitamins, minerals, herbs and dietary supplements for 4 days, dietary instruction will be provided. Blood samples will be taken at screen for safety labs. On study days 5, 13 and 21 a spot urine will be collected and a 7 hr serial blood draw will be performed at 0 hr, 30 min, 1 hr, 2 hr, 3 hr, 4 hr and 6 hr. Subjects will be provided with a light lunch with foods low in polyphenols. Subjects will only be able to eat the foods provided on the intervention days. Subjects will be asked to drink 32oz of water during the 7-hr period. Subjects will also be asked to collect all of their urines for 24 hrs, 2 consecutive days.
  Interventions: Dietary Supplement: Pomegranate Juice; Dietary Supplement: Soybean Flour Protein
- Soy Isolate Protein (Active Comparator): Subjects will be asked to take a dietary supplement on the day of intervention. Prior to intervention, subjects will be asked to avoid high-polyphenol foods, certain vitamins, minerals, herbs and dietary supplements for 4 days, dietary instruction will be provided. Blood samples will be taken at screen for safety labs. On study days 5, 13 and 21 a spot urine will be collected and a 7 hr serial blood draw will be performed at 0 hr, 30 min, 1 hr, 2 hr, 3 hr, 4 hr and 6 hr. Subjects will be provided with a light lunch with foods low in polyphenols. Subjects will only be able to eat the foods provided on the intervention days. Subjects will be asked to drink 32oz of water during the 7-hr period. Subjects will also be asked to collect all of their urines for 24 hrs, 2 consecutive days.
  Interventions: Dietary Supplement: Pomegranate Juice; Dietary Supplement: Soy Isolate Protein

INTERVENTIONS:
Dietary Supplement: Pomegranate Juice — Pomegranate Juice alone
Dietary Supplement: Soybean Flour Protein — Soybean Flour Protein combined with Pomegranate Juice
  Other Names: Nutrasorb
  Arms: Soybean Flour Protein
Dietary Supplement: Soy Isolate Protein — Soy Isolate Protein combined with Pomegranate Juice
  Other Names: Solae
  Arms: Soy Isolate Protein

SUMMARY:
This study is comparing the quantity of active metabolites from consuming pomegranate juice in three different preparations. People who participate in this study will come in to the Center for a screening visit, which includes a blood test and medical history. If you qualify based on the screening visit, you will then come in to the Center while fasting in the morning on three different days. You will eat a standardized breakfast and drink one of three juices, and then remain for metabolic testing at the Center for a period of time after eating. You will also be provided a standardized lunch and water during this period. Each of those visits will last about 7 hours. During this time, and for the rest of the 24 hours following drinking the juice, you will collect all of your urine. Following all three of these 7-hour visits, you will return to the Center again the next day for a fasting blood draw, drop off your urine sample, and pick up a new container to collect another 24 hour urine sample. The following day, you will return to the Center to drop off your second urine sample collection.

DETAILED DESCRIPTION:
Pomegranate (Punica granatum L.) fruits are widely consumed as pomegranate juice (PJ), and their health benefits have been studied extensively in animals and humans (1-6). The pomegranate fruit is a rich source of polyphenols, most of which are ellagitannins (ETs). Pomegranate extracts,which incorporate these major polyphenols from the pomegranate fruit, have been developed in dry and liquid forms to provide alternative convenient sources for obtaining the bioactive polyphenols found in PJ. We have previously reported on the pharmacokinetics and metabolism of pomegranate polyphenols, after the consumption of PJ in normal healthy human volunteers (7). In humans, ETs are converted to ellagic acid (EA) in the small intestines and absorbed with a maximum plasma concentration observed at approximately 1 hour. EA disappears from plasma 6 hours after administration of PJ. Ellagitannins and ellagic acid remaining in the intestine and are then further converted by gut microflora to urolithin-A, absorbed and derivatives, which are metabolized by phase II enzymes and excreted in human urine for up to 48 hours after consumption of PJ(7).

Polyphenols are dietary constituents of plants associated with health-promoting effects. In the human diet, polyphenols are generally consumed in foods along with macronutrients. Because the health benefits of polyphenols are critically determined by their bioavailability, the effect of interactions between plant phenols and food macronutrients is a very important topic. The protein-polyphenol complexes can significantly change the plasma kinetics profile. (8) Protein-polyphenol binding is mediated by a combination of hydrogen and hydrophobic bonding depending on chemical (polarity) and structural (size/shape) properties of interacting molecules. Covalent interactions between purified glycinin, a soybean storage protein, and selected flavonoids and phenolic acids have also been reported. Recently it is reported that protein-rich defatted soybean flour protects anthocyanins during transit through upper digestive tract for subsequent colonic delivery/metabolism (9).

ELIGIBILITY:
Inclusion Criteria:

* Male or female >20 and < 45 years of age at the time the consent form is signed.
* Subject must sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or randomization. A subject will be excluded for any condition that might compromise the ability to give truly informed consent for participation in the study.

Exclusion Criteria:

* Any subject who is eating more than 4 servings per day of fruits and vegetables, taking vitamin supplements or taking any antibiotics or other medication or dietary supplement which interfere with the absorption of polyphenols.
* Any subjects with a history of gastrointestinal surgery (except for appendectomy), diabetes mellitus, or other serious medical condition, such as chronic hepatitis or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as BP >160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease corrected with medication to normal laboratory values) as indicated by medical history or routine physical examination.
* Major surgery within 12 weeks prior to subject randomization and/or screening, especially cardiac surgery
* Is currently a smoker who has a therapeutic plan to quit smoking anytime during the study period; or if not a current smoker, has quit smoking within the past 3 months.
* Known HIV positive.
* Clinical evidence of current malignancy with the exception of basal cell or squamous cell carcinoma of the skin and cervical intraepithelial neoplasia.
* Currently receiving systemic chemotherapy and/or radiotherapy.
* Active bleeding.
* Subject has any disorder (excluding illiteracy or visual impairment) that compromises the ability of the subject to give written informed consent and/or to comply with study procedures.
* Subject who is allergic to soy protein.
* In the opinion of the study investigator has a risk of non-compliance with study procedures, or can not read, understand or complete study related materials.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 08/01/2014 - 01/31/2015. Enrollment took place in a private setting in the clinic located at the site.
Pre-assignment Details: After a 4-day washout period, participants received pomegranate juice (PJ) alone, PJ mixed with soy protein, or PJ mixed with soybean flour in random sequence with a 7-day washout in between.
Groups:
- PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein: Participants consumed PJ alone, then PJ+ soybean flour, then PJ + soy protein with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
- PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour: Participants consumed PJ alone, then PJ+ soy protein, then PJ + soybean flour with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
- PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein: Participants consumed PJ+soybean flour, then PJ alone, then PJ+soy protein with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
- PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ: Participants consumed PJ+soybean flour, then PJ+soy protein, then PJ alone with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
- PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ: Participants consumed PJ+soy protein, then PJ+soybean flour, then PJ alone with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
- PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour: Participants consumed PJ+soy protein, then PJ alone, then PJ+soybean flour with PJ dosing 236.5 mL, soy protein 20 g and soybean flour 20 g
Period: First Intervention (1 Day)
Arm/Group | PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein | PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour | PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein | PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ | PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ | PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein | PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour | PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein | PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ | PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ | PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein | PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour | PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein | PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ | PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ | PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein | PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour | PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein | PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ | PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ | PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | PJ First, Then PJ With Soybean Flour, Then PJ With Soy Protein | PJ First, Then PJ With Soy Protein, Then PJ With Soybean Flour | PJ With Soybean Flour First, Then PJ, Then PJ With Soy Protein | PJ With Soybean Flour First, Then PJ With Soy Protein, Then PJ | PJ With Soy Protein First, Then PJ With Soybean Flour, Then PJ | PJ With Soy Protein First, Then PJ, Then PJ With Soybean Flour
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since this was a crossover study, the total number of participants was 18 in each arm.
Groups:
- All Study Participants: Participants took pomegranate juice (PJ, 236.5 mL or 8 fl.oz) alone, or PJ (236.5 mL) mixed with 20 g of soy protein, or PJ (236.5 mL) mixed with 20 g of soybean flour in random order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Ellagic Acid Concentration 0 to 24 Hours Post-dose Area Under the Curve
Description: Blood samples were collected at baseline, 0.5, 1, 2, 3, 4, 6 and 24 h after ingestion of pomegranate juice (PJ) alone, or PJ mixed with soy protein, or PJ mixed with soybean flour. Plasma concentration of ellagic acid at each time point was determined to create a pharmacokinetic parameter area under the curve.
Time Frame: Baseline, 0.5, 1, 2, 3, 4, 6 and 24 hr after 1 dosing of each intervention during the 3-week period
Population: All participants for whom plasma ellagic acid was determined at baseline, 0.5, 1, 2, 3, 4, 6 and 24 hr after 1 dosing of PJ, or PJ with soy protein, or PJ with soybean flour
Measure: Mean (Standard Deviation); unit: micromol*h/L
Groups:
- All Study Participants Consuming PJ: Participants consumed PJ (236.5 mL) only
- All Study Participants Comsuming PJ With Soy Protein: Participants consumed PJ (236.5 mL) mixed with soy protein isolate (20 g)
- All Study Participants Comsuming PJ With Soybean Flour: Participants consumed PJ (236.5 mL) with soybean flour protein (20 g)
Arm/Group | All Study Participants Consuming PJ | All Study Participants Comsuming PJ With Soy Protein | All Study Participants Comsuming PJ With Soybean Flour
Number analyzed (Participants) | 18 | 18 | 0
micromol*h/L | 0.074 (0.029) | 0.075 (0.028) |
Statistical Analysis 1: Comparison: All Study Participants Consuming PJ vs All Study Participants Comsuming PJ With Soy Protein; Comparison of ellagic acid concentration 0 to 24 hours post-dose area under the curve was made to PJ alone vs. PJ with soy protein after intervention. Due to the quality issue of soybean flour, data from this intervention group was not analyzed; Test type: Other; p = 0.82, t-test, 2 sided; Mean Difference (Final Values) = 0.001

ADVERSE EVENTS:
Time Frame: Adverse data was collected over a 3 week period
Description: Participants were monitored and questioned regarding the occurrence and nature of any adverse experiences.
Groups:
- Study Participants Consuming PJ Alone: All participants consumed PJ (236.5 mL or 8 fl.oz) alone
- Study Participants Consuming PJ With Soy Protein: All participants consumed PJ (236.5 mL) mixed with 20 g of soy protein
- Study Participants Consuming PJ With Soybean Flour: All participants consumed PJ (236.5 mL) mixed with 20 g of soybean flour
Arm/Group | Study Participants Consuming PJ Alone | Study Participants Consuming PJ With Soy Protein | Study Participants Consuming PJ With Soybean Flour
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No